CLINICAL TRIAL: NCT02955719
Title: CAMH - McMaster Collaborative Care Initiative For Mental Health Risk Factors In Dementia: Depression, Anxiety, and Mild Cognitive Impairment
Brief Title: CAMH - McMaster Collaborative Care Initiative For Mental Health Risk Factors In Dementia
Acronym: CCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Tarek Rajji, Dr., Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 019/2016
Record Dates: First submitted 2016-10-24; First posted 2016-11-04 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Depression; Anxiety; Mild Cognitive Impairment
Keywords: Collaborative Care; Depression; Anxiety; Mild Cognitive Impairment; Integrated Care Pathway
MeSH Terms: conditions — Depression; Anxiety Disorders; Cognitive Dysfunction | interventions — Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enrolled Cases (Experimental): Integrated Care Pathway with different treatment interventions
  Interventions include:
  Sertraline, Venlafaxine, CBT/Psychological therapy, Psychiatric consultation, lifestyle intervention resources
  Interventions: Drug: Sertraline; Drug: Venlafaxine; Other: CBT/Psychological Therapy; Other: Psychiatric Consultation; Other: Lifestyle Intervention Resources
- Enrolled Controls (No Intervention): No intervention: Treatment as usual (TAU) will be provided by the primary care practice staff

INTERVENTIONS:
Drug: Sertraline
  Other Names: zoloft
  Arms: Enrolled Cases
Drug: Venlafaxine
  Other Names: effexor
  Arms: Enrolled Cases
Other: CBT/Psychological Therapy
  Arms: Enrolled Cases
Other: Psychiatric Consultation
  Arms: Enrolled Cases
Other: Lifestyle Intervention Resources
  Arms: Enrolled Cases

SUMMARY:
Age remains the single most significant risk factor for developing dementia, particularly Alzheimer's dementia (AD). Given the rate at which Canada's population is aging, the quest to determine modifiable risk factors, whether by prevention, earlier detection, or an ability to slow the rate of decline, is a key priority in health care. Primary care is likely to play a pivotal role in this initiative. Collaborative mental health care between primary care providers and mental health clinicians has been demonstrated to be effective at the patient and system levels. Thus, the overall goal of this project is to assess impact and feasibility of implementing a collaborative care evidence-based Integrated Care Pathway (ICP) in addressing three potentially reversible risk factors at high risk for developing AD: anxiety, depression, or mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The investigators will enroll 150 participants overall (CAMH and McMaster). Seventy-five will be cases who will be enrolled into the ICP arm of the study and these will be patients born in the calendar year 1951, 1953 or 1955. The investigators will enroll an additional 75 controls that were born in the calendar year 1950, 1952 or 1956.

Patients of general practitioners being seen at primary healthcare clinics in the Greater Toronto Area and in Hamilton, who were born in the calendar year 1950, 1951, 1952, 1953, 1955, or 1956 will be consented and screened for anxiety, depression, and Mild Cognitive Impairment (MCI).

If patients born in 1951, 1953 and 1955 reach a threshold level of anxiety, depression, or MCI symptom burden and have a confirmed diagnosis, rather than receive treatment as usual, the participants will be enrolled into an Integrated Care Pathway (ICP), which offers evidence-informed treatment for the management of these syndromes in a routine, algorithmic fashion. All enrolled cases entered in the study will be provided with general interventions that address lifestyle and medical factors that both contribute to these syndromes and are thought to predispose patients to develop dementia. If the symptom burden is severe enough, based on standardized assessments, evidence-based psychopharmacology (a trial of sertraline and/or venlafaxine) will also be offered, with a standardized titration schedule. Collaboration will be built into the ICP - a psychiatrist will be present at the clinic and in contact with primary care providers to provide patient- and physician-level support, consultation, and episodes of care as necessary. Rates of anxiety, depression, and MCI diagnosis/detection, time to treatment initiation, and improvement in symptom burden will be assessed.

If patients born in 1950, 1952 and 1956 reach a threshold level of anxiety, depression, or MCI symptom burden, these individuals will form our comparison group and will receive treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria

1. Female or male primary practice patients of participating physicians born in 1951, 1953 or 1955 (ICP) and 1950, 1952 or 1956 (TAU).
2. Can read and understand English.
3. Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.
4. Willing and able to provide informed consent

Exclusion Criteria:

1. Diagnosis of dementia.
2. Substance abuse identified as an acute problem in the four weeks before being enrolled in the study (i.e. the day the patient signs the informed consent form).
3. Those with delirium, or where we are unable to make a diagnosis of MCI, due to unstable comorbidities.
4. Palliative-care patients.

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Change in anxiety/depression/quality of life (QOL) scores among participants in the ICP and comparison groups | From Baseline Screening to 24 month follow-up
  Comparison for the GAD-7/PHQ-9/QOL scores will be assessed using Group x Time ANOVAs repeated measure comparing scores at assessment times in the intervention and comparison groups.

SECONDARY OUTCOMES:
Acceptability and perceived utility of the ICP | Baseline to 24 month follow-up
  Qualitative data will be gathered from primary care teams to determine the acceptability and perceived utility data from brief team meetings and focus groups.
Feasibility of the ICP | Baseline to 24 month follow-up
  Qualitative data for the feasibility indicators will be obtained from the information collected by the research coordinator from the primary care team during the recruitment, screening, and data collection phases of the study, as well as the chart review.
Adjustments made for the adoption of the ICP in primary care teams | Baseline to 24 month follow-up
  Qualitative data about the adjustments made at each primary care practice to adopt the ICP will be gathered from brief meetings and focus groups.
Barriers to implementation of the ICP and the key elements to initiate, sustain and spread the ICP | Baseline to 24 month follow-up
  Qualitative data on difficulties with implementing the ICP, as well as information on successfully initiating and supporting the ICP will be gathered from brief meetings and focus groups
Changes in the primary care providers' knowledge of, and ability to recognize and manage, depression, anxiety, and MCI in older adults. | Baseline to 24 month follow-up
  Mean ratings on the Primary Care Team Questionnaire will be calculated at baseline and at the end of the study and compared using t-tests.
Time-to-treatment initiation among those in the ICP arm versus those in the comparison arm. | Baseline to 24 month followup
  The length of time from identification of anxiety, depression or MCI and the start of the ICP intervention (i.e., time-to-treatment initiation) will be calculated in days for patients in the intervention group and comparison group. The average length of time-to-treatment initiation will be calculated for each group and these means will be compared using a t-test.
Specific Aim 3a: To assess the impact of the ICP on the rates of diagnoses/detection among older patients with anxiety, depression, or MCI compared to before ICP implementation. | Calculate one year prior to the time of Site Initiation Visit for all recruiting sites.
  During the recruitment phase of the study, charts of patients born in 1950, 1954 will be reviewed to identify diagnosis of depression, anxiety and/or MCI prior to the implementation of the ICP. The period of data collection for this chart review is calculated as one year prior to the time of the SIV for all sites.
Specific Aim 3b: To assess the impact of ICP on rates of diagnoses/detection among patients of the same age cohort as our target ICP population, but not in our study sample. | Calculate the 6 month period prior to the last study assessment for a given recruitment site.
  We will review contamination effects by reviewing the charts of clinic patients born in 1954 and 1958 to identify the diagnosis/detection of depression, anxiety and/or MCI in the 6 month period prior to the last study assessment for a given recruitment site.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Rajji, MD, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kates N, Craven M; Collaborative Working Group of the College of Family Physicians of Canada, Canadian Psychiatric Association. Shared mental health care. Update from the Collaborative Working Group of the College of Family Physicians of Canada and the Canadian Psychiatric Association. Can Fam Physician. 2002 May;48:936. No abstract available. PMID 12053639
- See also: : Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research